CLINICAL TRIAL: NCT03129425
Title: Quasi-experimental Study With a Control Group to Evaluate a Multidisciplinary Psychoeducational Intervention on Coping Skills, Psychosocial Adaptation and Quality of Life in Parkinson's Disease Patients and Cares
Brief Title: Quasi-experimental Study With a Control Group to Evaluate a Psychoeducational Intervention in Parkinson's Disease Patients and Carers
Acronym: ReNACE-PD01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ReNACE-PD01
Record Dates: First submitted 2017-04-11; First posted 2017-04-26 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Parkinson Disease
Keywords: Patient; Caregiver; Coping; Psychosocial adaptation
MeSH Terms: conditions — Parkinson Disease | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Sessions in groups
  Interventions: Behavioral: ReNACE Psychoeducational Intervention
- Control group (Sham Comparator): Sessions in groups
  Interventions: Other: General Educational Program

INTERVENTIONS:
Behavioral: ReNACE Psychoeducational Intervention — 9 sessions in groups of 15-20 people at most so as to promote reflection and facilitate the interchange of opinions between participants about issues of interest from their day to day experience of coping with Parkinson's disease.
  Other Names: Experimental group
  Arms: Intervention group
Other: General Educational Program — 5 sessions in groups of 15-20 people
  Other Names: Control group
  Arms: Control group

SUMMARY:
The aim of this study is to evaluate the effects of a psychoeducational multidisciplinary intervention focusing on improving coping skills, the psychosocial adaptation to Parkinson's disease and the quality of life in patents and family carers in a Primary Care setting.

On the basis of previous research, the hypothesis we propose is that through the development of coping skills which will contribute to promoting a positive psychosocial adaptation to Parkinson' disease, the quality of life of the people with Parkinson's disease and their family carers will be improved. At the same time, it is predicted that, by incorporating this psychoeducational intervention into clinical practice, the patients and family caregivers will perceive a greater sense of normality in their lives, which will also promote compliance with drug treatments and promote healthy lifestyles. In the long-term, such an approach could have positive effects on the overall health of patients and their family carers.

This quasi-experimental study with control group and mixed methods was designed to evaluate the ReNACE psychoeducational intervention (ReNACE is the spanish acronym for the Research Programme and means Recovery, Normalisation, Acceptance and Living with Chronic illness). Based on the relevant study power calculations, 100 people with Parkinson's disease and 100 family carers will be recruited. Participants will be assigned to two groups. The intervention group will receive the ReNACE psychoeducational intervention. The control group will be given a general educational program. The study will be carried out in community-based health centers. The results obtained from the two groups will be evaluated at three time points: at baseline, immediately after the intervention and at 6 months after the intervention. The results will be measured with the following instruments: the Quality of Life Scale PDQ-39 (The 39-item Parkinson's Disease Questionnaire) for patients and the Quality of Life Scale for caregivers SQLC (Scale of Quality of Life of Caregivers) for family carers, and for patients and family carers the Psychosocial Adjustment to Illness Scale Self-report (PAIS-SR) and the Brief Cope Inventory. To determine the acceptability of the intervention, focus groups will be organized with some patients and family carers who have received the ReNACE intervention and also with the healthcare professionals involved in its development.

DETAILED DESCRIPTION:
Registry procedures

* Letters will be sent from the centers themselves to the homes of all the people diagnosed with Parkinson's disease who meet the inclusion criteria. The letters will contain information about the study and how to join the study, a stamped addressed envelope and the informed consent form. Those interested may sign up for the study by telephone, by sending a letter in a stamped addressed envelope (provided by the research team) or in person at the reception of the participating centers. Subsequently, a member of the research team will evaluate if the potential participants meet the inclusion criteria by means of a brief interview in the health center. Once it has been established that participants fulfill the inclusion criteria, they will be given a document with the dates of the sessions that they must attend.
* The healthcare professionals helping the participants in data collection will be blinded to intervention assignment. Two researchers will be in charge of data monitoring.
* Data will be compared with findings from papers.
* The sample size necessary to detect medium to large differences in the primary outcome of the project, quality of life, was calculated. The parameters used for the calculation of the sample size by group will be published in a paper.
* Analysis of quantitative data will be performed on an intention to treat basis and for that SPSS (Statistical Package for the Social Sciences) version 23.0 will be used. A descriptive analysis of the sociodemographic data will be made. For the quantitative variables, the means of central tendency and standard deviations will be calculated. Non-parametric tests (χ² tests) and parametric tests (paired student t tests) to compare patients with family members at each measurement points, unpaired student t tests to determine any significant differences between the two groups at baseline (Time 0) and the measurements at Time 1 and Time 2 will be used. Also, repeated measures of covariance (ANCOVA, analysis of covariance) will be used to compare differences between the two groups in the main variables.

ELIGIBILITY:
Inclusion Criteria:

* People with Parkinson's disease receiving care as outpatients in the designated centers in any stage of the disease (as determined by a researcher with the Hoehn & Yahr scale), residing at that time in Navarra, fluent in the speaking and understanding of the Spanish language, and with preserved cognitive ability.
* Family members/carers will be over the age of 18, living or maintaining a close relationship with a patient and actively collaborating in the care of the patient, currently residing in Navarra and fluent in the speaking and understanding of the Spanish language

Exclusion Criteria:

* People with Parkinson's disease and family members who do not wish to participate.
* People with Parkinson's disease and family members who do not meet the inclusion criteria because of any event during the study time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Quality of life at 9 weeks and 24 weeks (6 months) in patients with Parkinson's disease | Baseline, 9 weeks and 24 weeks
  The quality of life is measured by the PDQ-39 (the 39-item Parkinson's Disease Questionnaire)
Change from Baseline Quality of life at 9 weeks and 24 weeks (6 months) in family carers | Baseline, 9 weeks and 24 weeks
  The quality of life is measured by the SQLC (Scale of Quality of Life of Caregivers)

SECONDARY OUTCOMES:
Change from Baseline Coping at 9 weeks and 24 weeks (6 months) | Baseline, 9 weeks and 24 weeks
  The scale of Brief Cope for patients and family carers
Change from Baseline Psychosocial adaptation to illness at 9 weeks and 24 weeks (6 months) | Baseline, 9 weeks and 24 weeks
  The scale PAIS-SR for patients and family carers (PAIS-SR: the Psychosocial Adjustment to Illness Scale Self-report)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier Mata Rodríguez, Study Chair — Director Research Department (OTRI). University of Navarre.
Locations (1):
- Servicio Navarro de Salud-Osasunbidea, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No
Participant data from scales will not be shared with other researchers.

REFERENCES:
- [Derived] Navarta-Sanchez MV, Ursua ME, Riverol Fernandez M, Ambrosio L, Medina M, Diaz de Cerio S, Alvarez MJ, Senosiain JM, Gorraiz A, Caparros N, Anaut S, Martin-Lanas R, Recio M, Portillo MC. Implementation of a multidisciplinary psychoeducational intervention for Parkinson's disease patients and carers in the community: study protocol. BMC Fam Pract. 2018 Apr 5;19(1):45. doi: 10.1186/s12875-018-0730-9. PMID 29621985